CLINICAL TRIAL: NCT00543075
Title: A Phase I Pharmacokinetic Study of Genasense® in Subjects With Normal Renal Function and Mildly and Moderately Impaired Renal Function
Brief Title: Pharmacokinetic Study of Genasense in Subjects With Normal Renal Function, Mildly Impaired Renal Function, and Moderately Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genta Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GPK104
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2008-06

CONDITIONS: Normal Renal Function; Mildly Impaired Renal Function; Moderately Impaired Renal Function
Keywords: Renal Function; Adult; Genasense; oblimersen; G3139; Genta; Pharmacokinetics
MeSH Terms: interventions — oblimersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Genasense (oblimersen, G3139) — 3 mg/kg/day by intravenous infusion for up to 48 hours
  Other Names: Oblimersen; G3139

SUMMARY:
To characterize the pharmacokinetics of G3139 in subjects with normal, mildly impaired, and moderately impaired renal function who receive Genasense 3 mg/kg/day by continuous intravenous infusion for 2 days (48 hours).

ELIGIBILITY:
Key inclusion criteria:

* Age > 18 years
* Adequate organ function as determined < 7 days prior to starting study medication (except for renal function, as specified per protocol)
* Creatinine clearance > 80 mL/min based on the Cockcroft-Gault formula for subjects in Group 1; or 50 to less than or equal to 80 mL/min based on the Cockcroft-Gault formula and confirmed based on measured creatinine clearance for subjects in Group 2; or 30 to 49 mL/min based on the Cockcroft-Gault formula and confirmed based on measured creatinine clearance for subjects in Group 3

Key exclusion criteria:

* Significant medical disease
* Prior organ allograft
* Coexisting condition that would require the subject to continue therapy during the treatment (infusion) phase of the study with a drug known to alter renal function

Min Age: 18 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-05; Primary Completion 2007-11 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of oblimersen (G3139) | Up to 58 hours after start of Genasense infusion

CONTACTS AND LOCATIONS:
Overall Officials: Harry Alcorn, PharmD, Principal Investigator — Davita Clinical Research
Locations (1):
- DaVita Clinical Research, Minneapolis, Minnesota, United States